CLINICAL TRIAL: NCT04960839
Title: Phase II Multicenter Clinical Trial of Prophylactic Irradiation to the Contralateral Breast for Breast Cancer Patients With BRCA1, BRCA2 and PALB2 Deleterious Mutation
Brief Title: Prophylactic Irradiation to the Contralateral Breast for BCAs Patients
Acronym: PICB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019-228
Record Dates: First submitted 2020-05-12; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: BRCA1; BRCA2; PALB2; Deleterious mutation; Prophylactic irradiation; Contralateral breast cancer risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (No Intervention): Standard loco-regional treatment without prophylactic contralateral breast irradiation
- Prophylactic irradiation group (Experimental): Standard loco-regional treatment with prophylactic contralateral breast irradiation
  Interventions: Radiation: Prophylactic contralateral breast irradiation

INTERVENTIONS:
Radiation: Prophylactic contralateral breast irradiation — The whole contralateral breast will be irradiated once daily, 5 days a week, for 5-6 weeks, using 1.8-2 Gy/fx to a total dose of 45-50 Gy.
  Arms: Prophylactic irradiation group

SUMMARY:
Breast cancer is the most common cancer in women worldwide, with high mortality. About 5% to 10% of breast cancers are hereditary. Most inherited cases of breast cancer are associated with germline mutations in genes, such as BRCA1, BRCA2 and PALB2. The cumulative breast cancer risk for BRCA1, BRCA2 or PALB2 mutation carriers was high.

Besides the increased breast cancer risk for the inherited mutation carriers, the risk of subsequent contralateral breast cancer for the mutation carriers with breast cancer was also significantly increased. Contralateral prophylactic mastectomy was usually recommended to the breast cancer patients with BRCA mutation. However, many breast cancer patients refused the contralateral prophylactic mastectomy, due to the surgical injury, potential surgical complications, deleteriously affected body image and sexuality.

Solid evidence validated that radiotherapy after surgery resulted in a reduced local recurrence for three times lower than surgery alone. It is thought that radiation would eliminate the microscopic tumors which may already exist in the breast. Thus, we proposed that for the breast cancer patients with BRCA1, BRCA2 or PALB2 deleterious germline mutations, prophylactic irradiation to the contralateral breast may reduce the risk of subsequent contralateral breast cancer. And we would like to further compare the effect of prophylactic irradiation to the published data from traditional prophylactic contralateral mastectomy.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women worldwide, with high mortality. In the US in 2018, the number of estimated new cases of breast cancer accounted for 30% of all the new cancer cases in women, while the estimated deaths of breast cancer accounted for 14% of all new cancer deaths. In Chinese females, the most commonly diagnosed cancer was breast cancer, accounting for 19% of total cases. And breast cancer was the main 5 most common causes of cancer-related deaths in China.

About 5% to 10% of breast cancers are hereditary. Most inherited cases of breast cancer are associated with germline mutations in two genes: BRCA1 (BRCA1 DNA repair associated) and BRCA2 (BRCA2 DNA repair associated). The cumulative breast cancer risk for BRCA1 or BRCA2 mutation carriers at age 70 years reached as high as 50% in US population and 37% in Chinese population. Benefiting from the next generation sequencing technology, more inherited gene mutations were discovered. Among these new discovered susceptibility genes, PALB2 (Partner and localizer of BRCA2) was associated with high increased risks of breast cancer in both Chinese and US population.

Besides the increased breast cancer risk for the inherited mutation carriers, the risk of subsequent contralateral breast cancer for the mutation carriers with breast cancer was also significantly increased. For contralateral breast cancer in BRCA mutation carriers, the cumulative risk for 10 years after breast cancer diagnosis was as high as 25% and for 20 years reached to 40%, as compared 3% and 12% respectively in non-carriers. Contralateral prophylactic mastectomy was usually recommended to the breast cancer patients with BRCA mutation, as it can absolutely reduce the risk of contralateral primary cancer. However, many breast cancer patients refused the contralateral prophylactic mastectomy, due to the surgical injury, potential surgical complications, deleteriously affected body image and sexuality.

Solid evidence validated that radiotherapy after surgery resulted in a reduced local recurrence for three times lower than surgery alone. It is thought that radiation would eliminate the microscopic tumors which may already exist in the breast. Thus, we proposed that for the breast cancer patients with BRCA1, BRCA2 or PALB2 deleterious germline mutations, prophylactic irradiation to the contralateral breast may reduce the risk of subsequent contralateral breast cancer. And we would like to further compare the effect of prophylactic irradiation to the published data from traditional prophylactic contralateral mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, aged 30-70yrs, diagnosed with stage 0-III breast cancer (NCCN-Breast Cancer V2.2019), undergoing the lumpectomy or mastectomy no more than 1 year. ALND or SLNB should be carried out and the lymph node status should be known.
* Patients with a deleterious germline mutation of BRCA 1/2 or PALB2.
* The patients with no contraindictation for irradiation.
* The patients consent for prophylactic irradiation to the contralateral breast.
* The patient may receive any regimen of adjuvant, neoadjuvant chemotherapy, according to the treating physician. The radiation therapy should start at least 2 weeks after the completion of all the chemotherapy cycles.
* The patient may receive endocrine therapy before, during or after study entry.
* The patient may receive target therapy (Trastuzumab) before, during or after study entry.
* The patient must be eligible for MRI examination of the contralateral breast.
* The patient refused prophylactic contralateral mastectomy and oophorectomy.

Exclusion Criteria:

* Metastatic breast cancer.
* Past history of other cancer besides breast cancer
* Previous irradiation of the breast or chest wall, but not for breast cancer treatment
* Synchronous bilateral breast cancer
* Patients with active connective tissue diseases, pneumonia are excluded due to the potential risk of significant radiotherapeutic toxicity.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Contralateral breast cancer | up to 10 years
  The recurrence rate of contralateral breast cancer

SECONDARY OUTCOMES:
Overal survival | up to 10 years
  The length of time from either the date of diagnosis or the start of lumpectomy or mastectomy for primary breast cancer with or without prophylactic irradiation to the contralateral breast
Ipsilateral loco-regional recurrence | Every 3-6 months. Follow up will be continued until 10 years after lumpectomy or mastectomy for primary breast cancer.
  Reappearance of cancer in the ipsilateral preserved breast, chest wall, axillary or supraclavicular lymph nodes.
Distant metastasis | up to 10 years
  Breast cancer that has spread from the original (primary) breast cancer to distant organs or distant lymph nodes.
Short time adverse effects | 3 months since radiation treatment start
  Any short term adverse effects that related to prophylactic irradiation
Long time adverse effects | up to 10 years
  Any long term adverse effects that related to prophylactic irradiation

CONTACTS AND LOCATIONS:
Overall Officials: Peifen Fu, M.D., Principal Investigator — Department of Breast Surgery, The First Affiliated Hospital, College of Medicine, Zhejiang University; Wenjun Chen, M.D., Principal Investigator — Department of Surgical Oncology, Sir Run Run Shaw Hospital, Zhejiang University; Kejin Wu, M.D., Principal Investigator — Department of Breast Surgery, Obsterics and Gynecology Hospital of Fudan University; Xiaowen Ding, M.D., Principal Investigator — Department of Breast Surgery, Cancer Hospital of University of Chinese Academy of Sciences; Zhengkui Sun, Principal Investigator — Department of Breast Surgery, Jiangxi Provincial Cancer Hospital; Mikael Hartman, Principal Investigator — Department of Surgery, Yong Loo Lin School of Medicine, National University of Singapore; Yiding Chen, Principal Investigator — Department of Breast Surgery, The Second Affiliated Hospital, Zhejiang University School of Medicine; Jiaojiao Zhou, Principal Investigator — Departmen of Breast Surgery, The Second Affiliated Hospital, Zhejiang University School of Medicine; Kun Zhang, Principal Investigator — Departmen of Breast Surgery, The Second Affiliated Hospital, Zhejiang University School of Medicine; Wenhong Xu, Principal Investigator — Departmen of Radiology, The Second Affiliated Hospital, Zhejiang University School of Medicine; Zhibing Wu, Principal Investigator — Department of Oncology, Zhejiang Hospital
Locations (8):
- China (7):
  - Department of Breast Surgery, Jiangxi Provincial Cancer Hospital, Jiangxi, Jiangxi
  - Department of Breast Surgery, Obestrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Department of Breast Surgery, Cancer Hospital of University of Chinese Academy of Sciences, Hangzhou, Zhejiang
  - Department of Breast Surgery, the First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Department of Breast Surgery, the Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Department of Surgical Oncology, Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou, Zhejiang
  - Department of Oncology, Zhejiang Hospital, Hangzhou, Zhejiang
- Department of Breast Surgery, Yong Loo Lin School of Medicine, National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No